CLINICAL TRIAL: NCT00253461
Title: Positron Emission Tomography Using 11C Topotecan in Predicting Response to Treatment in Patients With Brain Metastases Due to Ovarian, Small Cell Lung, or Other Cancer
Brief Title: 11C Topotecan PET Imaging
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drugs unavailable:unable to make radioactive topotecan
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CWRU6Y02; P30CA043703 (NIH); CASE-CWRU-6Y02 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Metastatic Cancer; Ovarian Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; extensive stage small cell lung cancer; recurrent small cell lung cancer; unspecified adult solid tumor, protocol specific; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; tumors metastatic to brain
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Small Cell Lung Carcinoma; Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: computed tomography — Within 4 weeks after initial imaging, patients also undergo a CT scan.
Procedure: positron emission tomography — Phase I: IV over 10 minutes followed immediately by a 1-2 hour positron emission tomography (PET) scan.
  Phase II: fludeoxyglucose F 18 IV and, 1 hour later, undergo a PET scan.
Radiation: 11C topotecan — Phase I and II: IV over 10 minutes
Radiation: fludeoxyglucose F 18 — Phase II: fludeoxyglucose F 18 IV

SUMMARY:
RATIONALE: Diagnostic procedures, such as positron emission tomography (PET scan) using 11C topotecan, may help doctors predict a patient's response to treatment and help plan the best treatment.

PURPOSE: This phase I/II trial is studying how well a PET scan using 11C topotecan predicts response to treatment in patients with brain metastases due to ovarian, small cell lung, or other cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if tumor uptake of ^11C topotecan occurs quickly enough and at sufficient concentration to be measured immediately following infusion in patients with brain metastases secondary to ovarian cancer, small cell lung cancer, or other cancers.
* Determine, preliminarily, if ^11C imaging has potential to be an early predictor of response to topotecan therapy in these patients.

Secondary

* Determine the whole-body biodistribution of ^11C topotecan in these patients.

OUTLINE:

* Phase I: Patients receive ^11C topotecan IV over 10 minutes followed immediately by a 1-2 hour positron emission tomography (PET) scan. Within 4 weeks after initial imaging, patients also undergo a CT scan.
* Phase II: Patients receive ^11C topotecan and undergo imaging as in phase I. Patients also receive fludeoxyglucose F 18 IV and, 1 hour later, undergo a PET scan.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian cancer, small cell lung cancer, or other cancers

  * Metastatic brain disease
* Eligible for topotecan therapy
* Measurable disease by CT scan and/or MRI

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Not specified

Renal

* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Adequate end-organ function
* Able to tolerate lying on a radiology table for ≥ 1 hour
* No serious medical or psychiatric illness that would preclude study compliance or giving informed consent

PRIOR CONCURRENT THERAPY: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics on day of positron-emission tomography scan | Within 1 week of PET
Disease response | after 1-2 courses of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Muzic, PhD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States